CLINICAL TRIAL: NCT06229015
Title: Evaluation of an Online Tool (E-TOOL) in the Selection of Patients for Spinal Cord Stimulation for Chronic Pain
Brief Title: Evaluation of Online Tool (E-TOOL SCS) in Spinal Cord Stimulaion
Acronym: E-TOOLSCS
Status: Enrolling by invitation | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Collaborators: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Sponsor
Other Study IDs: 2506 CE
Record Dates: First submitted 2024-01-05; First posted 2024-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Failed Back Surgery Syndrome; Limb Ischemia; Neuropathic Pain; Complex Regional Pain Syndromes
Keywords: Spinal cord stimulation; SCS-E-TOOL; Chronic Pain Treatment
MeSH Terms: conditions — Failed Back Surgery Syndrome; Neuralgia; Complex Regional Pain Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This observational multicenter study aims to evaluate the reliability and validity of the e-tool for selecting patients eligible for SCS for chronic pain caused by one of the four etiologies listed above in the experience of daily clinical practice. The implantation procedure and devices used will be those used in the routine clinical practice of participating centers. Since the study is observational, the use of the e-tool will not replace the routine medical and psychological evaluation in participating centers before SCS implantation.

Study Objectives:

Primary Objective: Evaluate the degree of agreement/disagreement between the physicians opinion and the e-tool in selecting patients eligible for spinal cord stimulation for chronic pain. Endpoint: Calculation of the probability of disagreement (πD) between the e-tool and the physicians opinion regarding the appropriateness of the intervention.

Secondary Objective: Evaluate the ability of the e-tool to classify interventions defined as appropriate and highly likely to succeed; (scores 7-9) at 3 different time points: trial, 6-month follow-up, and 12-month follow-up. The proportion of interventions that were successful at the trial implantation in different time points will be compared with the proportion of interventions identified as appropriate and highly likely to succeed by the e-tool.

Study Period: 24 months. 12 months of enrollment + 12 months of follow-up. Subjects: Number of subjects to be included: at least 60 (total divided between the two centers)

Participating Centers:

* Pain Therapy Unit - ICSMaugeri, Pavia
* Anesthesia and Pain Therapy SD - Azienda Ospedaliero Universitaria Pisana Pisa

DETAILED DESCRIPTION:
Spinal Cord Stimulation (SCS) has been a therapy in the treatment of chronic pain for 50 years, particularly for patients resistant to conventional pharmacological treatment and other less complex invasive procedures. Over the years, various versions of guidelines have been established and drafted for the selection and clinical indications in which SCS therapy is most likely to be successful. The main clinical indications include:

* Chronic pain in the lumbar region and lower limbs, especially in patients who have undergone spine surgeries (Failed Back Surgery Syndrome, FBSS).
* Complex Regional Pain Syndrome (CRPS).
* Peripheral neuropathic pain.
* Ischemic pain in the limbs. In daily clinical practice, the heterogeneity of patients often makes it difficult to determine which patients are eligible for this treatment. A large number of clinical studies suggest that cognitive aspects and individual coping mechanisms in dealing with pain experiences impact treatment response. For this reason, international guidelines recommend that individuals considered for SCS should undergo a comprehensive psychological evaluation.

Recently, an online tool (SCS-e-tool) has been implemented for selecting patients eligible for SCS implantation. Developed by a team of experts in pain therapy with various clinical backgrounds, this tool is freely available online and can be used by healthcare professionals. It is designed to assist in evaluating a patients suitability for spinal cord stimulation and aid in making informed clinical decisions.

The SCS-e-tool takes into account various factors, including cognitive aspects and the patient pain management modalities. The goal is to provide a comprehensive and personalized assessment to identify patients who may benefit most from spinal cord stimulation therapy. This tool can be a valuable aid for healthcare professionals in the decision-making process regarding patient selection for SCS therapy.

It is important to note that, despite the utility of assessment tools, the final decision on a patient candidacy for spinal cord stimulation should be based on a comprehensive evaluation that includes clinical, psychological, and individual aspects of the patient.

The implementation of tools like the SCS-e-tool represents a step forward in the personalized approach to chronic pain management and the optimization of patient selection for specific therapies such as spinal cord stimulation.

Recently, an online tool (SCS-e-tool) has been implemented for the selection of patients eligible for SCS implantation, developed by a pool of experts in pain therapy with diverse clinical profiles. This tool, available online for free and built according to the RUAM method, allows the input of various clinical profiles with diagnostic, clinical, and psychological information and provides indications on the likelihood of SCS success and suggestions regarding the need for psycho-social support therapies in conjunction with neurostimulation.

The e-tool scores range from 1 to 9 and are divided as follows: 1-3 inappropriate intervention, 4-6 intervention with uncertain outcomes, 7-9 appropriate intervention with a high probability of success. The e-tool has a dual use for implanters and referrers. For both groups, the scope is similar, but perspectives differ: Referrers perspective: appropriateness in terms of referring a patient to consider SCS as the next step in chronic pain management. Implanter's perspective: appropriateness in terms of selecting a patient for SCS as the next step in chronic pain management.

ELIGIBILITY:
Inclusion Criteria:

* • Males and females aged between 18 and 85 years.

  * Patients with chronic pain and indication for implantation of a temporary neurostimulator for spinal cord stimulation testing.
  * Signed informed consent.

Exclusion Criteria:

* • Patients who, in the researcher's judgment, are unable to follow the protocol instructions.

  * Patients in presumed/confirmed pregnancy.
  * Contraindications to implantation.

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chronic pain afferent to pain therapy units in ICS Maugeri hospital Pavia or in University Hospital Pisa
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-07-13 (Actual); Primary Completion 2022-01-16 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Numerical rating scale | through study completion, an average of 1 year
  Numeric Rating Scale (NRS): a scale for pain intensity assessment useful for controlling therapies, clinical routine monitoring, and scientific studies. The result is the indication of pain intensity on a scale from 0 to 10, where 0 indicates no pain, and 10 indicates the maximum imaginable pain

SECONDARY OUTCOMES:
Evaluate the ability of the E-TOOL to classify interventions defined as appropriate and highly likely to succeed | perioperatively/periprocedurally
  The proportion of interventions that were successful at the trial implantation will be compared with the proportion of interventions identified as approprite and highly likely to success by the E-TOOL
Oswestry Disability Index | through study completion, an average of 1 year
  Oswestry Disability Index (ODI): a standardized tool for assessing the degree of disability reported by a patient and related to pain symptoms but also to other disabling conditions. It assesses the interference of disability with various aspects of daily life
European Quality of life, EuroQol | through study completion, an average of 1 year
  European Quality of Life, EuroQoL (EQ-5D-5L): a standardized tool that measures the health status of respondents and their quality of life, based on which it is possible to assess the health care provided, a technique, a technology
Patient global impression of change (PGIC) | through study completion, an average of 1 year"
  Patient global impression of change (PGIC) is a 7 point scale depicting a patient's rating of overall improvement, and reflects a patient's belief about the efficacy of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- ICSMaugeri Spa, Pavia, Italy